CLINICAL TRIAL: NCT05967819
Title: Independent and Synergistic Effects of Physical and Psychosocial Stress on Functional Hypothalamic Amenorrhea in Exercising Women
Brief Title: Effects of Physical and Psychosocial Stress on Functional Hypothalamic Amenorrhea in Exercising Women
Acronym: FHA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Colorado Springs (Other)
Responsible Party: Principal Investigator, Marissa Baranauskas, Assistant Professor, University of Colorado, Colorado Springs
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: CRCW FHA
Record Dates: First submitted 2023-07-21; First posted 2023-08-01 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Amenorrhea Secondary
Keywords: functional hypothalamic amenorrhea; menstrual cycle; female athlete
MeSH Terms: interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Participants will be asked to maintain their usual physical activity and lifestyle habits.
- Exercise Stress (Experimental): The duration of participant's weekly running or cycling mileage will be increased by 30% while intensity is maintained.
  Interventions: Behavioral: Exercise Stress
- Psychosocial Stress (Experimental): Participants will be asked to complete cognitive function tasks designed to be stressful while maintaining their usual physical activity habits.
  Interventions: Behavioral: Psychosocial Stress
- Exercise + Psychosocial Stress (Experimental): Participants will be asked to complete cognitive function tasks designed to be stressful while the duration of their weekly running or cycling mileage is increased by 30% and intensity maintained.
  Interventions: Behavioral: Exercise Stress; Behavioral: Psychosocial Stress

INTERVENTIONS:
Behavioral: Exercise Stress — Increased exercise volume
  Arms: Exercise + Psychosocial Stress; Exercise Stress
Behavioral: Psychosocial Stress — cognitive tasks
  Arms: Exercise + Psychosocial Stress; Psychosocial Stress

SUMMARY:
The goal of this clinical trial is to determine how changes in exercise and psychosocial stress may influence the risk of menstrual cycle irregularities in female runners and cyclists. The main questions it aims to answer are:

* Does the implementation of exercise or psychosocial stress effect circulating reproductive hormones (i.e., estradiol, progesterone, luteinizing hormone) and menstrual cycle length?
* Is there an additive effect of combined exercise and psychosocial on circulating reproductive hormones (i.e., estradiol, progesterone, luteinizing hormone) and menstrual cycle length?

Participants will be asked to do the following over the ~3 month enrollment period:

* attend a laboratory visit at the beginning and end of the study to have their resting metabolic rate, aerobic fitness, and body composition tested
* monitor their menstrual cycle length, daily perceived stress levels, physical activity, and diet each month
* provide several urine and saliva samples each month
* either maintain their usual physical activity and lifestyle habits (control group), increase the duration of their weekly running or cycling mileage by 30% (exercise stress group), complete cognitive function tasks designed to be stressful (psychosocial stress group), or increase the duration of their weekly running or cycling mileage by 30% and complete cognitive function tasks designed to be stressful (exercise + psychosocial stress group) during the final month of enrollment.

Researchers will compare control, exercise stress, psychosocial stress, and exercise + psychosocial stress groups to see if there is an effect on circulating reproductive hormones (i.e., estradiol, progesterone, luteinizing hormone) and menstrual cycle length.

ELIGIBILITY:
Inclusion Criteria:

* participates in structured running or cycling exercise for at least 30 minutes on 4 days per week or more
* have regular periods every 21 to 35 days
* have not used hormonal contraceptives for at least the past 6 months
* are not currently or trying to become pregnant or are breastfeeding, and have not been pregnant or breastfeeding for the past 12 months
* have never been diagnosed with a menstrual cycle disorder (e.g., menorrhagia, amenorrhea, dysmenorrhea, polycystic ovary syndrome [PCOS], endometriosis, premenstrual dysphoric disorder [PMDD], menstrual migraines, ovarian cancer, ovarian insufficiency, uterine or endometrial cancer)
* have never been diagnosed with a metabolic disease (e.g., hypothyroidism, hyperthyroidism, Cushing disease, Addison's disease, diabetes)

Exclusion Criteria:

* missing > 4 consecutive days of aerobic exercise (i.e., running, cycling, cross training) if assigned to the exercise intervention groups
* they indicate they "Could not participate at all due to a health problem" or have had to modify their exercise training, felt their injury, illness, or other health problem has affected their exercise performance, or experienced symptoms/ health complaints greater than "To a minor extent" on the Oslo Sports Trauma Research Center Questionnaire (exercise training intervention group)
* demonstrate clinical low energy availability as defined as energy availability <30 Kcal/kg fat free mass in the first two months of at-home monitoring
* report menstrual cycle lengths <21 days or >35 days in the first two months of at-home monitoring
* do not demonstrate an anticipated rise in progesterone levels during the latter half of their cycle and luteinizing hormone levels at mid-cycle compared to tests taken during the first few days after menses in the first two months of at-home monitoring
* begin taking a hormonal contraceptive
* become pregnant
* are diagnosed with a menstrual cycle disorder (e.g., menorrhagia, amenorrhea, dysmenorrhea, polycystic ovary syndrome [PCOS], endometriosis, premenstrual dysphoric disorder [PMDD], menstrual migraines, ovarian cancer, ovarian insufficiency, uterine or endometrial cancer)
* are diagnosed with a metabolic disease (e.g., hypothyroidism, hyperthyroidism, Cushing disease, Addison's disease, diabetes), 10) are diagnosed with a major cardiovascular disease, respiratory disease, or musculoskeletal injury
* are unable to follow instructions for any of the procedures

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-08-09 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Urinary estrone-3-glucuronide (E3G) | 3 months
  ng/mL
Urinary pregnanediol glucuronide (PdG) | 3 months
  ug/mL
Urinary luteinizing hormone (LH) | 3 months
  MIU/mL
Menstrual cycle length | 3 months
  days

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Colorado Springs, Colorado Springs, Colorado, United States

IPD SHARING:
Plan to Share IPD: No